CLINICAL TRIAL: NCT03988062
Title: Aneurysm Packing With the Expandable TrelliX Coil System - A Prospective Safety Study
Acronym: APEX-FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shape Memory Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD1003
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ruptured or Unruptured Cerebral Aneurysms
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- TrelliX Embolic Coil System (Experimental)
  Interventions: Device: TrelliX Embolic Coil System

INTERVENTIONS:
Device: TrelliX Embolic Coil System — Embolic coil with shape memory polymer

SUMMARY:
APEX-FIH is a first-in-human, open-label prospective multicenter study of the TrelliX Embolic Coil System for use in embolization of the medium to large, ruptured or unruptured cerebral aneurysms

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥18 and ≤80 years with a diagnosis of a ruptured or unruptured intracranial aneurysm judged suitable for selective endovascular treatment by coil occlusion during single procedure
* Aneurysm size [largest measurement from the cross sectional images to determine overall aneurysm size, not just the lumen) ≥5 mm and ≤16mm
* If ruptured aneurysm: either WFNS grade 1 or 2, or Hunt and Hess 1 or 2
* If unruptured aneurysm: Subject grade Modified Rankin Scale mRS 0 - 2
* Investigator plans to use ≥70% in volume TrelliX coils to fill target aneurysm

Exclusion Criteria:

* Prior treatment (surgical or endovascular) of the target aneurysm
* Planned treatment of multiple aneurysms in index procedure
* Planned use of other modified coils (Matrix, HydroCoil or fibered coils)
* Planned use of liquid embolic material
* Life expectancy less than 12 months
* Presence of arteriovenous malformation
* Fusiform, mycotic, traumatic, or tumoral aneurysms
* Intended or planned aneurysm treatment by parent vessel occlusion
* Clipping or endovascular treatment of another intracranial aneurysm performed within 30 days before or planned within 30 days following the index procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Safety - Serious adverse events | 30 days
  Rate of freedom from incidence of serious adverse events related to the study
Efficacy - Angiographic occlusion | Immediate
  Rate of angiographic occlusion based on Raymond-Ray grading scale [1 No filling of aneurysm neck or dome; 2 Residual filling of aneurysm neck, not dome; 3 Residual filling of aneurysm neck and dome (worst outcome)]
Efficacy - Angiographic occlusion | 6 months and 12 months
  Rate of angiographic occlusion based on Raymond-Ray grading scale [1 No filling of aneurysm neck or dome; 2 Residual filling of aneurysm neck, not dome; 3 Residual filling of aneurysm neck and dome (worst outcome)]

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Hospital Clínico Regional Guillermo Grant Benavente, Concepción
  - Instituto de Neurocirugía, Santiago

IPD SHARING:
Plan to Share IPD: No